CLINICAL TRIAL: NCT01186185
Title: Mineralocorticoid Treatment for Sudden Sensorineural Hearing Loss
Brief Title: Fludrocortisone for Sudden Hearing Loss
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI moved to new institution, unable to complete study
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00006240
Record Dates: First submitted 2010-08-19; First posted 2010-08-23 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Hearing Loss, Sensorineural
Keywords: sudden; sensorineural; hearing loss; fludrocortisone; mineralocorticoid; steroid
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss | interventions — Fludrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fludrocortisone (Experimental)
  Interventions: Drug: Fludrocortisone

INTERVENTIONS:
Drug: Fludrocortisone — Fludrocortisone 0.2 mg by mouth daily for 30 days

SUMMARY:
The standard of care treatment of sudden hearing loss uses a type of steroid called glucocorticoid. Examples of glucocorticoids are prednisone, methylprednisolone and dexamethasone. Not everybody recovers hearing with glucocorticoid treatment. Fludrocortisone is a different type of steroid called mineralocorticoid. Unlike glucocorticoids, which work by reducing inflammation, mineralocorticoids work by changing salt and fluid balance. In animal studies, fludrocortisone is at least as effective as glucocorticoid in preserving hearing. Fludrocortisone is not approved for the treatment of sudden hearing loss. The purpose of this study is to test whether fludrocortisone can treat sudden hearing loss.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Idiopathic sudden sensorineural hearing loss within 3 months
* Failure to recover hearing with glucocorticoid treatment or inability to tolerate glucocorticoid

Exclusion Criteria:

* Other diagnosis for the sudden hearing loss
* Concurrent systemic use of another steroid
* Hypersensitivity to fludrocortisone
* Systemic fungal infection
* Hypertension requiring two or more medications
* Pitting edema
* Cardiomegaly
* Congestive heart failure
* Electrolyte abnormality
* Concurrent use of barbiturates, phenytoin, fosphenytoin, rifampin, or rifapentine

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Hearing | At one month
  Hearing outcome will be determine by pure-tone and speech audiometry measured at the completion of a one-month course of treatment and compared with pre-treatment test results.

CONTACTS AND LOCATIONS:
Overall Officials: Anh Nguyen-Huynh, MD PhD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No